CLINICAL TRIAL: NCT01295970
Title: Feasibility of a Prospective, Randomized Trial Comparing Surgery Versus Radiosurgery for the Treatment of Single Brain Metastases
Brief Title: Surgery Versus Radiosurgery for the Treatment of Single Brain Metastases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 10-0486-C
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Patients With a Single Brain Metastasis
Keywords: Surgery of the brain; Radiosurgery; Brain Metastasis
MeSH Terms: conditions — Brain Neoplasms | interventions — Surgical Procedures, Operative; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiosurgery (SRS) (Active Comparator)
  Interventions: Procedure: Stereotactic Radiosurgery
- Surgery (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Prior to surgery, patients will have placement of scalp fiducials and undergo a contrast enhanced MRI scan. Once the patient is anesthetized or sedated, the head will be secured with a head frame and scalp fiducials will be registered to the stereotactic neuronavigation system. The tumor will then be resected and the patient will be taken to the recovery unit.
  Arms: Surgery
Procedure: Stereotactic Radiosurgery — This will be delivered using Gamma Knife technology. Patients randomized to this arm will be fitted with a stereotactic head-frame for stereotactic localization of brain metastases.
  Arms: Radiosurgery (SRS)

SUMMARY:
Usually the treatment of a single brain metastasis is surgery or Stereotactic Radiosurgery (SRS). Surgery involves resection of the brain tumor by means of an operation, whereas SRS is treatment consisting of highly focused radiation doses to the tumor. These two treatment modalities are both widely used, well established, and proven to improve survival, but so far, no study has been done to directly compare the efficacy of one over the other. Neither treatment in itself is considered to be experimental and both have been shown to provide benefits to patients with metastatic brain tumors. The aim of this study is to determine which two modalities are better for local control and improving quality of life.

Patients who consent to this study will be randomized to either receive surgery or Radiosurgery in the treatment of single brain metastases. The study seeks to recruit 12 patient to each group. Patients will be in this study for up to five years from the time of the treatment finished. This will include follow-up visits at 4 weeks after the procedure and then every 3 months after the procedure up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven malignancy (original biopsy is adequate as long as the brain imaging is consistent with brain metastases)
2. Patients > 18 years
3. A contrast-enhanced MRI demonstrating the presence a single brain metastases <3cm performed within one month prior to registration
4. Life expectancy > 3 months
5. RPA Class 1 and RPA Class 2 patients with stable primary disease
6. Patients must have normal organ and marrow function
7. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
8. ECOG Performance Status 0-2
9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Have tumor(s) in the midbrain, pons, or medulla, in eloquent cortex
2. Have tumors within 10 millimeters of the optic apparatus (nerves and chiasm) or the area postrema
3. Be poor operative candidates from an anesthetic point of view secondary to other major medical illnesses
4. Have a coagulopathy demonstrated by an abnormal prothrombin time, activated partial thromboplastin time, or thrombocytopenia (platelet count less that 150,000 platelets/mm3)
5. Have radiographic or cerebrospinal fluid specimen evidence of widespread leptomeningeal metastasis
6. Significant psychiatric impairments which, in the opinion of the investigators, will interfere with the proper administration or completion of the protocol
7. Acute or untreated infections (viral, bacterial or fungal)
8. Be prisoners or other institutionalized individuals
9. Have a diagnosis of germ cell tumor, lymphoma or small cell lung cancer 10.Concurrent chemotherapy or molecularly targeted anti-cancer therapy

11.Allergy to Gadolinium 12.Imminent brain herniation, massive peritumoural oedema or hydrocephalus 13.Have any metallic implant that would exclude the possibility of having a brain MRI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of accrual to a randomized trial of SRS vs Surgery in patients with single brain metastasis. | 2 years
To compare the incidence of recommendation for a second local therapeutic intervention to the treated metastasis at 1 year. | 2 years

SECONDARY OUTCOMES:
To compare overall survival between the two randomized cohorts. | 2 years
To compare local-recurrence-free survival between the two randomized cohorts. | 2 years
To compare CTCAE v 3.0 neurological outcomes | 2 years
To evaluate difference in neurocognitive outcomes | 2 years
To measure and compare quality of life | 2 years
To determine adverse effects attributable to local therapy | 2 years
To compare medication requirements in each cohorts (steroids, anticonvulsants) | 2 years
To explore potential predictive factors of outcomes | 2 years
To investigate potential biofluid and imaging biomarkers of response | 2 years
To compare ECOG performance status | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Zadeh, MD, Principal Investigator — University Health Network, Toronoto Western Hospital